CLINICAL TRIAL: NCT05008861
Title: Safety of Gut Microbiota Reconstruction Plus PD-1/PD-L1 Monoclonal Antibodies to Treat Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: Gut Microbiota Reconstruction for NSCLC Immunotherapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2021-179R
Record Dates: First submitted 2021-08-12; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Nivolumab; durvalumab; sintilimab; tislelizumab; camrelizumab; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT with anti-PD-1/PD-L1 treatment (Experimental)
  Interventions: Procedure: Capsulized Fecal Microbiota Transplant; Drug: Anti-programmed cell death protein 1/programmed death-ligand 1 monoclonal antibody; Drug: Platinum based chemotherapy

INTERVENTIONS:
Procedure: Capsulized Fecal Microbiota Transplant — Capsules contained washed fecal microbiota.
  Other Names: Capsulized FMT
Drug: Anti-programmed cell death protein 1/programmed death-ligand 1 monoclonal antibody — Standard dose of one of anti-PD-1/PD-L1 mAbs administered as a 1 hour infusion every 3 weeks.
  Other Names: Anti-PD-1/PD-L1 mAb; Anti-PD-1/PD-L1; Pembrolizumab; Nivolumab; Durvalumab; Sintilimab; Tislelizumab; Camrelizumab
Drug: Platinum based chemotherapy — Standard dose of Platinum based Chemotherapy every 3 weeks.
  Other Names: Platinum based Chemotherapy drugs

SUMMARY:
In this study, patients with locally advanced or metastatic NSCLC after first-line treatment with PD-1/PDL-1 monoclonal antibody will be treated with Gut Microbiota reconstruction(such as FMT) combined with PD-1/PDL-1 monoclonal antibody. We will evaluate the safety of FMT in the treatment of advanced NSCLC, and analyze the effect of FMT on intestinal flora and immunophenotype of patients.

ELIGIBILITY:
Inclusion Criteria:

1.Volunteer to participate in this trial, fully understand this trial, and sign the Informed Consent Form (ICF).

2.18-75 years old on the day of signing the ICF. 3.Locally advanced/metastatic non-small cell lung cancer diagnosed by histology or cytology. no epidermal growth factor receptor (EGFR) sensitive mutations, anaplastic lymphoma kinase (ALK) gene rearrangement, ROS Proto-oncogene 1 (ROS1) gene fusion.

4.Have stable disease (SD) defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 after receive at least 2 doses of anti-PD-1/PD-L1 for first-line treatment.

5.Have not received systemic treatment for locally advanced/metastatic NSCLC before immunotherapy.

6.Have measurable target lesions judged by the investigator according to Response Evaluation Criteria In Solid Tumors (RECIST V1.1).

7.0~1 ECOG score. 8.Life expectancy ≥ 12 weeks. 9.Have sufficient organ function, evaluated based on blood routine, renal function, liver function, and coagulation laboratory test results (and have not received blood transfusion or infusion of apheresis components within 14 days before the study drug administration , Erythropoietin, granulocyte colony stimulating factor and other medical support treatments).

10.Women of Childbearing Potential (WOBCP) must undergo a serum pregnancy test within 7 days before the first medication, and the result is negative; WOBCP or men and their WOBCP partners should agree from signing the ICF to the last one. Take effective contraceptive measures within 6 months after taking the study drug.

Exclusion Criteria:

1. Before the first administration of the anti-PD-1/PD-L1 reatment: a) have received previous systemic cytotoxic chemotherapy for metastatic disease; b) have received other targeted or biological anti-tumor therapy for metastatic disease ; c) received major surgery (<3 weeks before the first dose); d) received lung radiotherapy >30 Gy within 6 months before the first dose of the trial treatment; e) the first trial treatment Palliative radiotherapy was completed within 7 days before administration.
2. Any other form of anti-tumor therapy is expected during the study period.
3. Have progressive disease (PD) or response(CR or PR) defined by RECIST v1.1 after receive at least 2 doses of anti-PD-1/PD-L1 for first-line treatment.
4. Unable to tolerate anti-PD-1/PD-L1 treatment due to adverse events or other reasons.
5. Unable to swallow FMT capsules.
6. Received antibiotic treatment within 30 days before the planned FMT started.
7. Fecal occult blood test or calprotectin positive; have ulcerative colitis, Crohn's disease, ischemic enteritis, infectious enteritis, etc not suitable to take intestinal bacteria capsules, but not include anti-PD-1/PD-L1-related colitis.
8. Live virus vaccines have been vaccinated within 30 days before the planned treatment. Seasonal influenza vaccine without live virus is allowed.
9. A history of past malignant disease is known, unless the subject receives potentially curative treatment and there is no evidence of disease recurrence within 5 years after starting treatment.
10. Accompanying known active central nervous system (CNS) metastasis and/or cancerous meningitis.
11. According to the standard of Common Adverse Event Terminology (CTCAE) 4th edition, peripheral neuropathy has been ≥2 grade.
12. Severe hypersensitivity reactions to other monoclonal antibody treatments have occurred in the past.
13. Accompanied by active autoimmune diseases, systemic treatment (ie, use of disease modifiers, corticosteroids or immunosuppressive drugs) is required within the past 2 years.
14. Are receiving long-term systemic steroid therapy. Subjects with asthma who require intermittent use of bronchodilators, inhaled steroids, or topical steroid injections are not excluded.
15. Have received any other anti-PD-1 or PD-L1 or PD-L2 drugs or antibodies in the past, or small molecule therapy that targets other immunomodulatory receptors or mechanisms. Participated in any other anti-PD-1/PD-L1 trials and received anti-PD-1/PD-L1 treatment. Such antibodies include (but are not limited to) antibodies against IDO, PD-L1, IL-2R and GITR.
16. Active infections requiring treatment.
17. Known human immunodeficiency virus (HIV) history (known HIV1/2 antibody positive). Accompanied by known active hepatitis B or C.
18. Being pregnant or breastfeeding, or expecting to conceive or conceive during the period of study drug treatment and within the required contraceptive period after the last administration of the study drug.
19. The researcher believes that there are any circumstances that are not suitable for selection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of FMT-related Adverse Events | 2 years
  Number of patients with adverse events after FMT
Incidence of anti-PD-1/PD-L1-related Adverse Events | 2 years
  Number of patients with adverse events related to anti-PD-1/PD-L1 after FMT

SECONDARY OUTCOMES:
Changes in diversity and composition of gut microbiota | 2 years
  Compare the difference of gut microbiota diversity and composition between pre-FMT and post-FMT samples. Microbiota diversity will be quantified by α-diversity ( Faith's Phylogenetic Diversity) based on meta-genomics sequencing. Microbiota composition will be quantified by the operational taxonomic unit (OTU) in the stool.
Efficiency of FMT engraftment | 2 years
  Evaluate the acquired similarity of the recipient microbiota to the donor microbiota by measuring the Euclidian distance between donor microbial composition and every available time point of the corresponding recipients, starting from the pre-FMT sample.
Changes in concentration of peripheral blood mononuclear cells | 2 years
  Compare composition and content of peripheral blood mononuclear cells (CD8+T-cells, NK cells and myelin-sourced inhibitory cells) between pre-FMT and post-FMT samples. The composition and content of CD8+T-cells, NK cells and myelin-sourced inhibitory cells were analyzed by flow cytometry.
Changes in concentration of tumor immune related cytokines | 2 years
  Compare the contents of tumor immune related cytokines (IFNγ、TNF、Granzyme A/B、Perforin and et al) between pre-FMT and post-FMT samples. The contents of tumor immune related cytokines were analyzed by enzyme-linked immunosorbent assay.
Objective response rate (ORR) | 2 years
  Number of patients with objective responses divided by the total number of evaluable patients, according to imaging studies (RECIST 1.1) and iRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Xizhong Shen, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Yes
  Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be available from the principal investigator Taotao Liu at shen.xizhong@zs-hospital.sh.cn, beginning 6 months and ending 5 years after the trial results were published. The study protocol and statistical analysis plan are available online from https://clinicaltrials.gov/. All proposals requesting data access will need to specify how it is planned to use the data, and all proposals will need approval of all investigators before data release.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months and ending 5 years after the trial results were published.
Access Criteria: All proposals requesting data access will need to specify how it is planned to use the data, and all proposals will need approval of all investigators before data release.
URL: http://clinicaltrials.gov/